CLINICAL TRIAL: NCT00130013
Title: Comparison of Standard Versus Double Dose of Amoxicillin in the Treatment of Non-Severe Pneumonia in Children Aged 2-59 Months: A Multi-Centre Randomized Double Blind Controlled Trial in Pakistan
Brief Title: Efficacy of Single Versus Double Dose of Oral Amoxicillin for Non-Severe Pneumonia in Children
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: ARI Research Cell (Other Government)
Collaborators: World Health Organization (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DDoseAmoxy
Record Dates: First submitted 2005-08-12; First posted 2005-08-15 (Estimated); Last update posted 2005-09-23 (Estimated); Status verified 2004-07

CONDITIONS: Pneumonia
Keywords: Children; Non-severe pneumonia; Oral amoxicillin
MeSH Terms: conditions — Pneumonia | interventions — Amoxicillin

INTERVENTIONS:
Drug: Oral Amoxicillin

SUMMARY:
The World Health Organization's (WHO) standard case management strategy for reducing acute respiratory infection (ARI) related mortality recommends oral cotrimoxazole and oral amoxicillin as first line drugs for the treatment of pneumonia. In 1989, the Pakistan Ministry of Health (MOH) adopted this strategy to control ARI mortality and recommended cotrimoxazole for treatment of outpatients pneumonia due to lower costs. A number of studies subsequently performed have shown significant in vivo and in vitro resistance of H. influenzae and S. pneumoniae, the commonest bacteria causing childhood pneumonia, to cotrimoxazole.

Although on a case by case basis for pneumonia, in vitro resistance does not correlate very well with in vivo failures, nevertheless, clinical failure rate for pneumonia therapy has increased in Pakistan over the years. One can hypothesize that if bacterial pneumonia is a certain proportion of all pneumonia cases, the rise in clinical failures may be related to increasing antimicrobial resistance. Therefore, it is probable that this rising clinical failure rate could be a reflection of increasing resistance. There may be an increase in antimicrobial resistance of S. pneumoniae and H. influenzae to amoxicillin over the period of years and the rising treatment failure could be a reflection of the rising minimum inhibitory concentrations (MIC's) (> 2 mcg/ml for H. influenzae, 1993-94), thereby, resulting in this increasing failure rate.

For the current study the researchers propose a multicentre, randomized, controlled double blind trial in which standard versus double dose oral amoxicillin for three days for the treatment of non-severe pneumonia in children less than five years of age will be compared.

Primary Objective:

To compare the proportion of children 2 - 59 months of age presenting with non-severe pneumonia, who achieve clinical resolution on day 5 with standard (15 mg/kg/8hrly) versus double dose (30 mg/kg/8hrly) of oral amoxicillin therapy given for 3 days.

Secondary Objective:

To follow the clinical course of non-severe pneumonia with the alternative criteria of treatment failure (signs of deterioration i.e. lower chest indrawing and appearance of danger signs) on or before day 3 and compare them with other children who have persistent fast breathing (respiratory rate above the cut off for age) on day 3.

Hypothesis:

Therapy outcome with double dose of oral amoxicillin is not different than the standard dose of amoxicillin, when used for three days for the treatment of non-severe pneumonia in 2-59 months old children.

DETAILED DESCRIPTION:
INTRODUCTION:

World Health Organization's (WHO) standard case management strategy for reducing ARI related mortality recommends oral cotrimoxazole and oral amoxicillin as first line drugs for the treatment of pneumonia. In 1989, the Pakistan Ministry of Health (MOH) adopted this strategy to control ARI mortality and recommended cotrimoxazole for treatment of outpatients pneumonia due to lower costs. A number of studies subsequently performed have shown significant in vivo and in vitro resistance of H. influenzae and S. pneumoniae, the commonest bacteria causing childhood pneumonia, to cotrimoxazole.

This increase in clinical failure with oral cotrimoxazole has put a lot of pressure both at national and international forums on the National ARI Control Programme of Pakistan to change its recommendations from cotrimoxazole to amoxicillin as the first line of therapy. Besides being efficacious for non-severe pneumonia amoxicillin has shown good efficacy in children with severe pneumonia and bacteremic children.

Although on a case by case basis for pneumonia, in vitro resistance does not correlate very well with in vivo failures, one can hypothesize that if bacterial pneumonia is a certain proportion of all pneumonia cases, the rise in clinical failures may be related to increasing antimicrobial resistance of S. pneumoniae and H. influenzae to amoxicillin.

It is felt that WHO criteria for treatment failure are too stringent. Improvement is defined as the return of respiratory rate to below the cut off for that particular age at 48 hours. Some of the children with viral pneumonia will continue to have respiratory rate above the cut off on the first follow-up. These children are otherwise well and show no signs of deterioration of the disease but according to WHO criteria they would be classified as treatment failure. The treatment failure rates hence are influenced by the definitions used.

The existing data shows that if the dose of amoxicillin is increased to achieve higher MICs, then the eradication of causative organism tend to be much more complete. As yet, no clinical trial has been conducted to address this important question in the treatment of childhood pneumonia.

The researchers propose a multicentre, randomized, controlled double blind trial in which standard versus double dose oral amoxicillin for three days for the treatment of non-severe pneumonia in children less than five years of age will be compared.

Primary Objectives:

1. To compare the proportion of children 2 - 59 months of age presenting with non-severe pneumonia, who achieve clinical resolution on day 5 with standard (15 mg/kg/8hrly) versus double dose (30 mg/kg/8hrly) of oral amoxicillin therapy given for 3 days.

Secondary Objective:

To follow the clinical course of non-severe pneumonia with the alternative criteria of treatment failure (signs of deterioration i.e. lower chest indrawing and appearance of danger signs) on or before day 3 and compare them with other children who have persistent fast breathing (respiratory rate above the cut off for age) on day 3.

Null Hypothesis:

Therapy outcome with double dose of oral amoxicillin is not different than the standard dose of amoxicillin, when used for three days for the treatment of non-severe pneumonia in 2-59 months old children.

STUDY POPULATION AND SITE:

Patients:

They will be recruited from those coming to outpatient departments (OPD) in large tertiary care hospitals in Pakistan.

CONSENT:

The purpose of the study will be explained to parents and oral informed consent to participate obtained.

Laboratory Workup:

Chest radiographs will be taken for all enrolled patients.

Study Design:

This will be a randomized, double blind, multi-centre trial.

Definitions:

ARI is defined according to the WHO ARI Programme guidelines 2 for children who have either a cough or difficult breathing.

A clinical resolution is defined as return of respiratory rate to normal (no pneumonia) according to WHO ARI standard case management classification 2.

Clinical Failure is defined as development of chest indrawing; or any other danger sign; or persistence of fast breathing at day 5 follow-up or thereafter leading to therapy change.

Improved will be defined as slower respiratory rate (either back to normal range for age, or lower by more than 5 compared to previous evaluation), feeding better according to mother and lower body temperature than previous assessment.

Same will be defined as still breathing fast (respiratory rate ± 5 breaths/minute compared to previous evaluation or higher than that), with no chest indrawing and or danger sign.

Worse will be defined as development of lower chest indrawing or any danger sign.

A relapse is defined as development of recurrence signs of pneumonia till day 14 after fast breathing has disappeared initially.

Follow-up:

All children will be followed-up on day 3, 5 and 14.

Sample size:

Keeping in mind the overall treatment failure rate of 20.9% with amoxicillin from the MASCOT study (1999 - 2001), it is expected that the proportion of patients who will fail to respond with standard dose amoxicillin will be around 21.0%.7 In order for double dose to be more efficacious there should be a difference of more than 5% in the treatment success rate as compared to the standard dose. The researchers assume that the failure rate will not be more than 13% with double dose amoxicillin. By using the power of 80% and the confidence interval of 95%, the estimated sample size comes to 369 for each group. Assuming the loss to follow up to be 15% (as it is an out patient study and having day 14 follow-up) the estimated sample size will be 425 patients in each group, a total of 850 patients. Thus 900 patients will be enrolled in one and a half ARI season.

ADVERSE REACTIONS:

Antibiotics such as amoxicillin are generally well tolerated and are rarely associated with serious or life threatening adverse reactions (possibly or probably related to drug therapy). The most common side effects reported include:

Allergic - skin rash, hives, itching or wheezing Digestive - nausea, vomiting, diarrhea Metabolic - moderate or transient increase in liver function tests - transaminases Hematological - anemia, leucopenia and irreversible thrombocytopenia

Rare side effects include anaphylactic shock, Stevens- Johnson syndrome and pseudomembranous colitis.

Identifying, managing and reporting adverse events:

The site investigator will carefully monitor each child for adverse events. If an adverse event occurs, the site investigator will assess its duration, seriousness, intensity and relationship to the duration of study medication (amoxicillin). The principal investigator will use their judgement about whether to continue the child in the study or to discontinue enrollment. The event and its treatment will be noted on appropriate CRFs and reported to the DSMC.

DATA ENTRY AND ANALYSIS:

Data forms will all be filled on auto copy forms and will be reviewed by the site co-ordinator.

Data will be entered using Epi Info 6 and will be entered twice by two separate operators and both data bases will be validated using Epi Info 6.

Outcome measures:

A clinical resolution is defined as return of respiratory rate to normal (no pneumonia) on day 5, according to WHO ARI standard case management classification.

Clinical/treatment Failure is defined as development of chest indrawing; or any other danger sign; or persistence of fast breathing at day 5 follow-up or thereafter leading to therapy change.

Data analysis:

Analysis will be carried out on intention to treat basis. For primary outcome proportion of therapy failures and their 95% CI will be calculated for both the two regimens. Then the researchers will compare proportion of therapy failure using alternative criteria and WHO defined conventional therapy failure criteria.

ELIGIBILITY:
Inclusion Criteria:

* They are aged 2-59 months.
* Diagnosed with WHO defined non-severe pneumonia

Exclusion Criteria:

* Children with signs of WHO defined severe or very severe disease.
* Known penicillin allergy, with a history of accelerated rash, urticaria, or anaphylactic symptoms. Complicating acute non-pulmonary or chronic illness.
* The children living outside the municipal limits of the city who cannot be followed up.
* Children who have taken the appropriate doses of WHO-recommended dose of antimicrobial drug for 48 hours prior to presentation.
* Children who have prior history of wheezing or bronchial asthma and are wheezing now.
* Children whose parents or guardians refuse to give consent.
* Previously enrolled patients in the present study.
* Hospitalization in the past two weeks.

Ages: 2 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 900
Dates: Start 2003-09; Study Completion 2004-06

PRIMARY OUTCOMES:
To compare standard vs double dose of oral amoxicillin for non-severe pneumonia in children < 5 age.

SECONDARY OUTCOMES:
To use modified treatment failure criteria on or before day 3 and compare them with WHO criteria for failure.

CONTACTS AND LOCATIONS:
Overall Officials: Tabish Hazir, Fellowship, Principal Investigator — ARI Research Cell, Children Hospital, Pakistan Institute of Medical Sciences, Islamabad, Pakistan
Locations (1):
- ARI Research Cell, Children Hospital, Pakistan Institute of Medical Sciences, Islamabad, Capital, Pakistan